CLINICAL TRIAL: NCT05519592
Title: Proximal Lower Limb Intramuscular Block : Effects on Hemiparetic Gait
Acronym: ProxiBlock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, ETIENNE SAVARD, Hospital Practictioner, Henri Mondor University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2022-A01457-36
Record Dates: First submitted 2022-08-19; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Neurologic Disorder; Spastic Hemiplegia; Gait, Hemiplegic; Block
MeSH Terms: conditions — Nervous System Diseases; Hemiplegia; Gait Disorders, Neurologic; Bites and Stings | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine (Experimental): Ropivacaine intramuscular injection
  Interventions: Drug: Ropivacaine injection
- Control (Placebo Comparator): Sodium Chlorure intramuscular injection
  Interventions: Drug: Sodium Chloride Injection

INTERVENTIONS:
Drug: Ropivacaine injection — Intramuscular ropivacaine injection (gluteus maximus and rectus femoris)
  Arms: Ropivacaine
Drug: Sodium Chloride Injection — Intramuscular sodium chloride injection (gluteus maximus and rectus femoris)
  Arms: Control

SUMMARY:
To assess feasability, tolerance of anesthesic intramuscular motor block. To study immediate effects on differents muscles : gluteus maximus, rectus femoris in a hemiparetic population (over 15 days) To precise the role of the muscles which could be rehabilitatoin targets.

DETAILED DESCRIPTION:
Spastic paresis comprises both muscular and neurological disorders affecting movement through mostly the antagonist muscles compared to the agonist : muscular : spastic myopathy, shortening, stretch-sensitive paresis and neurogenic : spastic dystonia and cocontraction.

About gait, most of the litterature focuses on distal muscles targets. There are no studies about proxmial muscles role (gluteus maximus). Anesthesic perineural block have the disavantage to induce sensitive block as intramuscular block do not.

ELIGIBILITY:
Inclusion Criteria:

* able to consent
* avoiding ground swing phase gait disorder

Exclusion Criteria:

* severe cognitive disorder
* INR > 3.5
* local cutaneous affection on injection sites
* acute medical affection
* seizure
* hypersensitivity to anesthesics
* brugada syndrome
* porphyria
* severe cardiac disorder
* polyradiculopathy
* botulinum toxin injection < 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-09 (Estimated); Primary Completion 2023-05-02 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the active amplitude of hip flexion, knee flexion and ankle flexion | baseline, day 7 and day 14

SECONDARY OUTCOMES:
change from baseline of the walking speed, at maximal speed, with shoes | baseline, day 7 and day 14
change from baseline of the walking speed, at maximal speed, without shoes | baseline, day 7 and day 14
change from baseline of the walking speed, at comfortable speed with shoes | baseline, day 7 and day 14
change from baseline of the walking speed, at comfortable speed without shoes | baseline, day 7 and day 14
change from baseline of the right step length, at maximal speed, with shoes | baseline, day 7 and day 14
change from baseline of the left step length, at maximal speed, with shoes | baseline, day 7 and day 14
change from baseline of the left step length, at maximal speed, without shoes | baseline, day 7 and day 14
change from baseline of the right step length, at maximal speed, without shoes | baseline, day 7 and day 14
change from baseline of the right step length, at comfortable speed, without shoes | baseline, day 7 and day 14
change from baseline of the right step length, at comfortable speed, with shoes | baseline, day 7 and day 14
change from baseline of the left step length, at comfortable speed, with shoes | baseline, day 7 and day 14
change from baseline of the left step length, at comfortable speed, without shoes | baseline, day 7 and day 14
change from baseline of the cadence (step per second), at comfortable speed, without shoes | baseline, day 7 and day 14
change from baseline of the cadence (step per second), at comfortable speed, with shoes | baseline, day 7 and day 14
change from baseline of the cadence (step per second), at maximal speed, with shoes | baseline, day 7 and day 14
change from baseline of the cadence (step per second), at maximal speed, without shoes | baseline, day 7 and day 14
change from baseline of Proprioception detection of gluteus maximus (minimal detectable change in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Proprioception detection of hamstrings (minimal detectable change in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Proprioception detection of vastus (minimal detectable change in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Proprioception detection of rectus femoris (minimal detectable change in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Proprioception detection of soleus (minimal detectable change in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Proprioception detection of gastrocnemius (minimal detectable change in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Passive range of motion of gluteus maximus (muscle length in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Passive range of motion of rectus femoris (muscle length in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Passive range of motion of vastus (muscle length in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Passive range of motion of soleus (muscle length in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Passive range of motion of gastrocnemius (muscle length in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of Passive range of motion of hamstrings (muscle length in degrees) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of spasticity (angle in degrees) of hamstrings | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of spasticity (angle in degrees) of gluteus maximus | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of spasticity (angle in degrees) of rectus femoris | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of spasticity (angle in degrees) of vastus | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of spasticity (angle in degrees) of soleus | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of spasticity (angle in degrees) of gastrocnemius | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of active amplitude against gastrocnemius | baseline, day 7 and day 14
change from baseline of active amplitude against soleus | baseline, day 7 and day 14
change from baseline of active amplitude against hamstrings | baseline, day 7 and day 14
change from baseline of active amplitude against gluteus maximus | baseline, day 7 and day 14
change from baseline of active amplitude against rectus femoris | baseline, day 7 and day 14
change from baseline of active amplitude against vastus | baseline, day 7 and day 14
change from baseline of fatigability against vastus (in degrees, after 15 second of alternative movement) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of fatigability against rectus femoris (in degrees, after 15 second of alternative movement) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of fatigability against gluteus maximus (in degrees, after 15 second of alternative movement) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of fatigability against hamstrings (in degrees, after 15 second of alternative movement) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of fatigability against gastrocnemius (in degrees, after 15 second of alternative movement) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of fatigability against soleus (in degrees, after 15 second of alternative movement) | baseline, day 7 and day 14
  using the five steps assessment (Gracies JM)
change from baseline of patient global impression of improvement | baseline, day 7 and day 14
  GPI-I questionnaire
change from baseline of right foot pressure distribution | baseline, day 7 and day 14
change from baseline of left foot pressure distribution | baseline, day 7 and day 14
change from baseline of left foot load | baseline, day 7 and day 14
change from baseline of right foot load | baseline, day 7 and day 14
change from baseline of stride velocity variability | baseline, day 7 and day 14
change from baseline of stride length variability | baseline, day 7 and day 14
change from baseline of stride time variability | baseline, day 7 and day 14
change from baseline of stance time variability | baseline, day 7 and day 14
change from baseline of double support time variability | baseline, day 7 and day 14
change from baseline of swing time assymetry | baseline, day 7 and day 14
change from baseline of stride time assymetry | baseline, day 7 and day 14
change from baseline of stride time | baseline, day 7 and day 14
change from baseline of swing time | baseline, day 7 and day 14
change from baseline of stance time | baseline, day 7 and day 14
change from baseline of stride velocity | baseline, day 7 and day 14

IPD SHARING:
Plan to Share IPD: Undecided